CLINICAL TRIAL: NCT01544361
Title: A Phase 1, Randomized, Placebo-controlled, Single-dose Study to Evaluate the Safety of MEDI7814 in Adult Volunteers
Brief Title: A Phase 1 Study to Evaluate the Safety of MEDI7814 in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CD-RI-MEDI7814-1027
Record Dates: First submitted 2012-02-15; First posted 2012-03-05 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: Healthy subjects; MEDI7814; FTiH

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): A single dose of placebo matched to MEDI7814 intravenous infusion over at least 60 minutes on Day 1.
  Interventions: Other: Placebo
- MEDI7814, 1 MG/KG (Experimental): A single dose of MEDI7814, 1 milligram per kilogram (mg/kg) intravenous infusion over at least 60 minutes on Day 1.
  Interventions: Biological: MEDI7814, 1 MG/KG
- MEDI7814, 3 MG/KG (Experimental): A single dose of MEDI7814, 3 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Interventions: Biological: MEDI7814, 3 MG/KG
- MEDI7814, 10 MG/KG (Experimental): A single dose of MEDI7814, 10 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Interventions: Biological: MEDI7814, 10 MG/KG
- MEDI7814, 20 MG/KG (Experimental): A single dose of MEDI7814, 20 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Interventions: Biological: MEDI7814, 20 MG/KG

INTERVENTIONS:
Other: Placebo — A single dose of placebo matched to MEDI7814 intravenous infusion over at least 60 minutes on Day 1.
  Arms: Placebo
Biological: MEDI7814, 1 MG/KG — A single dose of MEDI7814, 1 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Arms: MEDI7814, 1 MG/KG
Biological: MEDI7814, 3 MG/KG — A single dose of MEDI7814, 3 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Arms: MEDI7814, 3 MG/KG
Biological: MEDI7814, 10 MG/KG — A single dose of MEDI7814, 10 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Arms: MEDI7814, 10 MG/KG
Biological: MEDI7814, 20 MG/KG — A single dose of MEDI7814, 20 mg/kg intravenous infusion over at least 60 minutes on Day 1.
  Arms: MEDI7814, 20 MG/KG

SUMMARY:
This is a Phase 1 study to evaluate the safety and tolerability of single ascending intravenous doses of MEDI7814 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of single ascending intravenous doses of MEDI7814 in healthy adult male subjects and female subjects of non-childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years up to and including 49 years at the time of first dose of investigational product
* Healthy by medical history, physical examination, and laboratory studies
* Body weight 50-125 kilogram (kg); body mass index 19.0-32.0 kilogram per square meter (kg/m^2) (inclusive)
* Females must be of non-childbearing potential.

Exclusion criteria:

* Any acute illness within 30 days of screening
* Concurrent enrollment in another clinical trial
* The subject has a positive drug/alcohol screen at screening or Day -1
* Pregnancy
* Current cigarette smokers
* History of cancer other than non-melanoma skin cancer or in situ carcinoma of the cervix treated with apparent success
* Use of immunosuppressive medications
* Subjects who have an unresolved infection with any Neisseria species
* Subjects who have had their spleen removed for any reason.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Marion, MD, Principal Investigator — Research site
Locations (1):
- Research Site, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 125 participants enrolled, 32 participants were randomized to treatment.
Period: Overall Study
Arm/Group | Placebo | MEDI7814, 1 MG/KG | MEDI7814, 3 MG/KG | MEDI7814, 10 MG/KG | MEDI7814, 20 MG/KG
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Placebo | MEDI7814, 1 MG/KG | MEDI7814, 3 MG/KG | MEDI7814, 10 MG/KG | MEDI7814, 20 MG/KG | TOTAL
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (9.9) | 28.5 (6.8) | 36.5 (6.7) | 28.0 (8.9) | 42.8 (4.0) | 33.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 4 | 7
  Male | 6 | 6 | 5 | 6 | 2 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study drug and up to Day 106 that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Day 1 to Day 106
Population: Safety population included all randomized participants who received MEDI7814 and had safety data available.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI7814, 1 MG/KG | MEDI7814, 3 MG/KG | MEDI7814, 10 MG/KG | MEDI7814, 20 MG/KG
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants
  TEAEs | 4 | 2 | 4 | 3 | 1
  SAEs | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetic (PK) Parameters of MEDI7814
Description: Individual MEDI7814 plasma concentration data and descriptive statistics of the PK parameters were to be tabulated by treatment group. Non-compartmental PK data analysis were to be performed for MEDI7814-treated participants to estimate PK parameters if data allowed.
Time Frame: Predose, end of infusion, 2, 6, 12 hours post-end of infusion on Day 1; Day 2, 3, 5, 8, 15, 22, 29, 43, 57, 85, and 106
Population: Analyses of PK was not performed as the clinical development of MEDI7814 had been discontinued because the indication was no longer being pursued.
Arm/Group | Placebo | MEDI7814, 1 MG/KG | MEDI7814, 3 MG/KG | MEDI7814, 10 MG/KG | MEDI7814, 20 MG/KG
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) for MEDI7814
Time Frame: Day 1, 29, 57, 85, and 106
Population: Analyses of immunogenicity was not performed as the clinical development of MEDI7814 had been discontinued because the indication was no longer being pursued.
Arm/Group | Placebo | MEDI7814, 1 MG/KG | MEDI7814, 3 MG/KG | MEDI7814, 10 MG/KG | MEDI7814, 20 MG/KG
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 106
Arm/Group | Placebo | MEDI7814, 1 MG/KG | MEDI7814, 3 MG/KG | MEDI7814, 10 MG/KG | MEDI7814, 20 MG/KG
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/8 | 2/6 | 4/6 | 3/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | MEDI7814, 1 MG/KG (N=6) | MEDI7814, 3 MG/KG (N=6) | MEDI7814, 10 MG/KG (N=6) | MEDI7814, 20 MG/KG (N=6)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | MEDI7814, 1 MG/KG (N=6) | MEDI7814, 3 MG/KG (N=6) | MEDI7814, 10 MG/KG (N=6) | MEDI7814, 20 MG/KG (N=6)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Analyses of PK parameters and immunogenicity were not performed as the clinical development of MEDI7814 had been discontinued because the indication was no longer being pursued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.